CLINICAL TRIAL: NCT04443413
Title: A Phase III Trial of Hypofractionated Radiotherapy to the Whole Breast or Post-Mastectomy Chest Wall Including Regional Nodal Irradiation
Brief Title: Phase III Study of 5tx vs 15tx of RT (X-rays or Protons) Including RNI in Breast Cancer Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MC1935; NCI-2020-04328 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1935 (Other: Mayo Clinic in Arizona); 19-008858 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8
MeSH Terms: interventions — Proton Therapy; Protons; X-Ray Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Panel-assessed cosmetic outcome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (x-ray therapy) (Experimental): Within 12 weeks of the last breast cancer surgery or last dose of adjuvant chemotherapy and no sooner than 14 days since the last chemotherapy, patients undergo x-ray therapy over 25 fractions in the absence of disease progression or unacceptable toxicity. Optionally, patients may then receive a 4-fraction boost of x-ray therapy.
  Interventions: Other: Questionnaire Administration; Radiation: X-ray Therapy
- Arm II (proton beam radiation therapy) (Experimental): Within 12 weeks of the last breast cancer surgery or last dose of adjuvant chemotherapy and no sooner than 14 days since the last chemotherapy, patients undergo proton beam radiation therapy over 5 fractions in the absence of disease progression or unacceptable toxicity. Optionally, patients may receive a concurrent 5-fraction boost of proton beam radiation therapy.
  Interventions: Radiation: Proton Beam Radiation Therapy; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: Proton Beam Radiation Therapy — Undergo proton beam radiation therapy
  Other Names: PBRT; Proton; Proton EBRT; Proton External Beam Radiotherapy; Proton Radiation Therapy; PROTON Therapy; Radiation, Proton Beam; External beam radiation therapy protons (procedure); External Beam Radiotherapy (protons)
  Arms: Arm II (proton beam radiation therapy)
Other: Questionnaire Administration — Ancillary studies
Radiation: X-ray Therapy — Undergo x-ray therapy
  Other Names: X-ray Radiation Therapy
  Arms: Arm I (x-ray therapy)

SUMMARY:
This phase III trial compares the rate of complications of x-ray therapy versus proton beam radiation therapy after breast conserving surgery or mastectomy in treating patients with breast cancer. X-ray therapy is a form of radiation therapy that uses high-energy radiation from x-rays to kill tumor cells and shrink tumors. Proton beam radiation therapy is a type of radiation therapy that uses high-energy beams to treat tumors. It is not yet known what level of complications x-ray therapy or proton beam radiation therapy have in treating patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the 24-month complication rate of 5 fraction radiotherapy compared to 25 fraction radiotherapy.

SECONDARY OBJECTIVES:

I. To evaluate acute toxicity that occur up to 12 months after radiation. II. To evaluate late toxicity that appear or persist 12 months after radiation. III. To estimate the 5-year locoregional control, invasive disease-free survival, disease-free survival, cause-specific survival and overall survival.

CORRELATIVE AND EXPLORATORY OBJECTIVES:

I. To evaluate patient-reported quality of life outcomes through Mayo Breast Survey, Mayo 10 (Patient-Reported Outcomes [PRO]-Common Terminology Criteria for Adverse Events [CTCAE]), and Mayo Patient Survey.

II. To evaluate clinical features, treatment technique, dose-volume parameters, histologic and genetic variants associated with fair and poor cosmetic outcomes or unplanned surgical intervention.

III. To evaluate the costs and comparative effectiveness of treatment. IV. Compare the use of photon therapy with spot scanning proton therapy hypo-fractionated whole breast or post-mastectomy chest wall with regional nodal irradiation.

V. To evaluated cosmetic outcome with patient-reported measures with elements from the Mayo Breast Patient Survey and panel assess cosmetic outcome with blinded photographs, and the Harvard/National Surgical Adjuvant Breast and Bowel Project (NSABP)/Radiation Therapy Oncology Group (RTOG) Cosmesis Scale.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Within 12 weeks of the last breast cancer surgery or last dose of adjuvant chemotherapy and no sooner than 14 days since the last chemotherapy, patients undergo x-ray therapy over 25 fractions in the absence of disease progression or unacceptable toxicity. Optionally, patients may then receive a 4-fraction boost of x-ray therapy.

ARM II: Within 12 weeks of the last breast cancer surgery or last dose of adjuvant chemotherapy and no sooner than 14 days since the last chemotherapy, patients undergo proton beam radiation therapy over 5 fractions in the absence of disease progression or unacceptable toxicity. Optionally, patients may receive a concurrent 5-fraction boost of proton beam radiation therapy.

After completion of study treatment, patients are followed up at 12 weeks, at 6, 12, 24, and 36 months, and then at 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological confirmation of breast cancer
* Breast conserving surgery or mastectomy (reconstruction is allowed)
* Clinical or pathologic T1-T4c, N0-3, M0 disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 2
* Able to and provides Institutional Review Board (IRB) approved study specific written informed consent
* Indications for breast or post mastectomy radiation with regional nodal radiotherapy per the discretion of the treating physician
* If uncertain of eligibility please consult the principal investigator (PI)

Exclusion Criteria:

* Medical contraindication to receipt of radiotherapy
* Severe active co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator or PI, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or providing informed consent
* Active systemic lupus or scleroderma
* Prior receipt of ipsilateral breast or chest wall radiation
* Persistent positive margins on ink after definitive surgery either for ductal carcinoma in situ (DCIS) or invasive cancer
* No active metastatic disease from other origin
* Recurrent breast cancer
* Patient requires bilateral breast radiation treatment
* cT4d patients (inflammatory breast cancer)
* Patients that may not be compliant or fit for the study at the discretion of the PI
* Male patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2026-11-19 (Estimated); Study Completion 2029-11-19 (Estimated)

PRIMARY OUTCOMES:
Complication rate | At 24 months
  Will be defined as the percentage of women evaluable at 24 months who develop one or more of these events: grade 3 or higher late adverse event or unplanned surgeries for cosmetic or treatment related events, including surgeries to remove implant.

SECONDARY OUTCOMES:
Incidence of acute adverse events | Up to 12 months post-radiation therapy
  The maximum grade for each type of acute adverse event will be recorded for each patient. Data will be summarized as frequencies and relative frequencies by treatment arm. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. Rates will be compared between arms using chi-squared tests.
Incidence of late toxicity | Up to 5 years post-radiation therapy
  Will be defined as any adverse event that occurred or persisted after the first 12 months post-radiation therapy and up to 5 years post-radiation therapy. The maximum grade for each type of late adverse event will be recorded for each patient. Data will be summarized as frequencies and relative frequencies by treatment arm. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. Rates will be compared between arms using chi-squared tests.
Locoregional control | Up to 5 years post-radiation therapy
  The cumulative incidence of locoregional recurrence will be estimated using a competing risks method by treatment arm. The competing risks will be distant breast cancer recurrence and death. Comparison between arms will employ Fine-Gray regression.
Invasive disease-free survival | From study registration until the time of invasive disease recurrence (not including ductal carcinoma in situ) or death due to any cause, assessed up to 5 years post-radiation therapy
  Invasive disease recurrence is defined by ipsilateral breast tumor recurrence (IBTR), regional recurrence, or distant recurrence. Will be estimated with a Kaplan-Meier estimator and curve by treatment arm. Estimates will be given for specific time points along with 95% confidence intervals. Comparison between arms will employ a log-rank test.
Disease-free survival | Up to 5 years post-radiation therapy
  Defined as the time from registration until the time of disease recurrence or death due to any cause. Will be estimated with a Kaplan-Meier estimator and curve by treatment arm. Estimates will be given for specific time points along with 95% confidence intervals. Comparison between arms will employ a log-rank test.
Cause-specific survival | Up to 5 years post-radiation therapy
  Will be estimated with a Kaplan-Meier estimator and curve by treatment arm. Estimates will be given for specific time points along with 95% confidence intervals. Comparison between arms will employ a log-rank test.
Overall survival | Up to 5 years post-radiation therapy
  Defined as the time from registration to death due to any cause. Will be estimated with a Kaplan-Meier estimator and curve by treatment arm. Estimates will be given for specific time points along with 95% confidence intervals. Comparison between arms will employ a log-rank test.

OTHER OUTCOMES:
Cosmetic outcome | Up to 5 years post-radiation therapy
  Will compare cosmetic outcome with patient self-reported and panel-assessed cosmetic outcome measures to include elements from the Mayo Breast Patient Survey, blinded photograph assessment, the modified Harvard/National Surgical Adjuvant Breast and Bowel Project/Radiation Therapy Oncology Group Cosmesis Scale, and the Breast Cancer Treatment Outcome Scale. Will be summarized with the frequencies and confidence intervals of fair or poor cosmesis events at baseline, 2 years, and 5 years by treatment arm. Comparisons between arms will employ chi-squared tests.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E. Vargas, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials